CLINICAL TRIAL: NCT05076344
Title: Understanding the Consequences of Recreational Noise Exposure
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: University of Manchester (Other); Nottingham University Hospitals NHS Trust (Other); National Institute for Health Research Nottingham Biomedical Research Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21021; MR/V01272X/1 (Other Grant/Funding Number: Medical Research Council (MRC) Programme Grant); 295085 (Other: IRAS Project ID); 21/LO/0615 (Other: Research Ethics Committee); 50341 (Other: Central Portfolio Management System (CPMS))
Record Dates: First submitted 2021-09-28; First posted 2021-10-13 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-03

CONDITIONS: Hearing Loss; Hearing Loss, Noise-Induced
Keywords: central nervous system; peripheral nervous system; magnetic resonance imaging
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Noise-Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1: young adults: 50 adults aged 18-19 years, with low lifetime noise exposure and audiometric thresholds in the normal range for their age.
- Group 2: older adults with low noise exposure: 50 adults aged 30-50 years, with low lifetime noise exposure and audiometric thresholds in the normal range for their age.
- Group 3: older adults with high noise exposure: 50 adults aged 30-50 years, with high lifetime noise exposure and audiometric thresholds in the normal range for their age.
- Group 4: older adults with suspected noise-induced hearing loss: 50 adults aged 30-50 years, with high lifetime noise exposure and audiometric thresholds above the normal range for their age.

SUMMARY:
The aim of this study is to determine whether measures derived from Magnetic Resonance Imaging (MRI) scans, and clinical and behavioural measures of hearing loss, in the peripheral and central auditory system (ranging from the cochlear nerve through the auditory brainstem to the auditory cortex) are associated with age and history of noise exposure in otherwise healthy adult humans.

DETAILED DESCRIPTION:
Noise exposure is the main cause of preventable hearing loss worldwide. Noise exposure occurs in the workplace, such as in noisy factories, and recreationally through the use of personal music players and attendance at nightclubs and live music events.

Hearing loss is usually diagnosed using pure tone audiometry, which measures the sensitivity of the ear to quiet sounds by determining the levels of tones that can just be heard at several test frequencies. Until recently, it had been assumed that hearing loss results mainly from damage to the sensory hair cells in the cochlea, the part of the ear that converts acoustic vibrations into electrical impulses in the cochlear nerve (CN). However, recent results from animal studies suggest that even moderate noise exposure can cause substantial damage to the CN, without any noticeable damage to the hair cells. Crucially, these results suggest that such damage does not immediately affect sensitivity to quiet sounds, but may exacerbate the effects of ageing.

Hearing loss is a huge problem. Substantial numbers of people, millions in the United Kingdom (UK) alone, are routinely exposed to significant levels of occupational and/or recreational noise. A large UK study found that one in seven adults aged 17-30 years reported "great difficulty" hearing speech in noisy backgrounds, while only one in fifty had impaired sensitivity as measured by pure tone audiometry. Hearing loss can lead to social isolation, depression, and is likely to be predictive of more severe hearing loss in old age. Recent studies suggest that hearing loss also reduces quality of life and is a risk factor for dementia.

This study is part of a programme grant conducted from April 2021 to March 2026 by The University of Manchester and The University of Nottingham. The overall aim of the programme is to understand the consequences of recreational noise exposure through improvement of the understanding of the contribution of CN damage to listening difficulties and audiometric losses.

The primary research questions are:

1. How does auditory pathway integrity vary with noise exposure, audiometric / outer hair cell (OHC) loss, and age?
2. How do auditory pathway integrity, audiometric loss, and OHC loss relate to listening difficulties? The secondary research question is to address how MRI measures relate to electrophysiological measures of auditory pathway integrity.

All participants will undergo the following non-invasive examinations:

* Extended high frequency audiometry to 16 kHz.
* Distortion Product Otoacoustic Emissions (DPOAEs): DPOAEs to 10.5 kHz.
* Middle Ear Muscle Reflex (MEMR): using a broadband contralateral elicitor and a click probe.
* Auditory Brainstem Response (ABR) to assess cochlear synaptopathy and central neural function. The ABR will be elicited with high-pass clicks.
* Speech in noise: A masked speech test will comprise verbal stimuli presented through headphones. The signal-to-background ratio will be varied adaptively to determine reception threshold.
* The Auditory Digit Span test to assess both forward and backward recall as a measurement of short term memory and working memory.
* The Tinnitus Functional Index to assess the severity of tinnitus.
* The Noise Exposure Structured Interview (NESI) to assess the lifetime noise exposure.
* MR Neurography using structural Magnetic Resonance Imaging to visualise the cochlear nerve and measure the diameter/cross-sectional area.
* High-resolution diffusion tensor imaging (DTI) to determine the apparent diffusion coefficient (ADC) and fractional anisotropy (FA) in the cochlear nerve.
* Whole-brain DTI to measure the apparent diffusion coefficient (ADC) and fractional anisotropy (FA) in the ascending auditory pathway and auditory cortex.
* High spatial resolution quantitative T1 mapping will be used to assess myelination in the ascending auditory pathway and auditory cortex.
* High spatial resolution T1 weighted imaging will be used to assess morphometry in the ascending auditory pathway and auditory cortex.
* Resting State Functional MRI, lasting 15 minutes, with eyes open and relaxed fixation, will be used to assess the functional connectivity in the ascending auditory pathway and auditory cortex.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent in English
* In the age range stipulated for the group, i.e. 18-19 inclusive for group 1 and 30-50 inclusive for groups 2 - 4.
* Audiometric thresholds in the range stipulated for the group, i.e. in the normal range for their age group for groups 1 - 3 and outside the normal range for their age group for group 4.
* Noise exposure in the range stipulated for the group, as determined by the NESI, i.e. less than 15 units for groups 1 - 2 and 15 or more units for groups 3 - 4.

Exclusion Criteria:

* Contraindications for MRI
* Motor impairment (for example, cerebral palsy)
* Cognitive impairment (for example, dementia or brain injury)
* Health conditions indicative of peripheral neuropathy (e.g. Type 1 diabetes).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals able to travel to the Sir Peter Mansfield Imaging Centre, University Park Campus of the University of Nottingham for up to three visits. Recruitment will be targeted to maximise the opportunities to recruit participants with noise exposure and suspected noise induced hearing loss.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Auditory nerve health | Baseline
  Auditory nerve diameter and/or surface area
Auditory nerve health | Baseline
  Diffusion measure in the auditory nerve (fractional anisotropy or apparent diffusion coefficient)

SECONDARY OUTCOMES:
Anatomical measure of the ascending auditory pathway | Baseline
  Diffusion measure in the ascending auditory pathway (fractional anisotropy or apparent diffusion coefficient)
Anatomical measure of the ascending auditory pathway | Baseline
  Myelination measure in the ascending auditory pathway
Anatomical measure of the ascending auditory pathway | Baseline
  Morphometry measure in the ascending auditory pathway
Functional measure of the ascending auditory pathway | Baseline
  Resting state functional connectivity measure in the ascending auditory pathway

CONTACTS AND LOCATIONS:
Overall Officials: Susan T Francis, PhD, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Hearing Theme, NIHR Nottingham Biomedical Research Centre, Ropewalk House, 113 The Ropewalk, Nottingham, Nottinghamshire
  - Sir Peter Mansfield Imaging Centre, University of Nottingham, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gates GA, Schmid P, Kujawa SG, Nam B, D'Agostino R. Longitudinal threshold changes in older men with audiometric notches. Hear Res. 2000 Mar;141(1-2):220-8. doi: 10.1016/s0378-5955(99)00223-3. PMID 10713509
- [Background] Kujawa SG, Liberman MC. Acceleration of age-related hearing loss by early noise exposure: evidence of a misspent youth. J Neurosci. 2006 Feb 15;26(7):2115-23. doi: 10.1523/JNEUROSCI.4985-05.2006. PMID 16481444
- [Background] Gopinath B, Schneider J, Rochtchina E, Leeder SR, Mitchell P. Association between age-related hearing loss and stroke in an older population. Stroke. 2009 Apr;40(4):1496-8. doi: 10.1161/STROKEAHA.108.535682. Epub 2009 Feb 26. PMID 19246693
- [Background] Deal JA, Albert MS, Arnold M, Bangdiwala SI, Chisolm T, Davis S, Eddins A, Glynn NW, Goman AM, Minotti M, Mosley T, Rebok GW, Reed N, Rodgers E, Sanchez V, Sharrett AR, Coresh J, Lin FR. A randomized feasibility pilot trial of hearing treatment for reducing cognitive decline: Results from the Aging and Cognitive Health Evaluation in Elders Pilot Study. Alzheimers Dement (N Y). 2017 Jun 21;3(3):410-415. doi: 10.1016/j.trci.2017.06.003. eCollection 2017 Sep. PMID 29067347
- [Background] Livingston G, Huntley J, Sommerlad A, Ames D, Ballard C, Banerjee S, Brayne C, Burns A, Cohen-Mansfield J, Cooper C, Costafreda SG, Dias A, Fox N, Gitlin LN, Howard R, Kales HC, Kivimaki M, Larson EB, Ogunniyi A, Orgeta V, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care: 2020 report of the Lancet Commission. Lancet. 2020 Aug 8;396(10248):413-446. doi: 10.1016/S0140-6736(20)30367-6. Epub 2020 Jul 30. No abstract available. PMID 32738937
- [Background] Guest H, Dewey RS, Plack CJ, Couth S, Prendergast G, Bakay W, Hall DA. The Noise Exposure Structured Interview (NESI): An Instrument for the Comprehensive Estimation of Lifetime Noise Exposure. Trends Hear. 2018 Jan-Dec;22:2331216518803213. doi: 10.1177/2331216518803213. PMID 30295145
- [Background] Meikle MB, Henry JA, Griest SE, Stewart BJ, Abrams HB, McArdle R, Myers PJ, Newman CW, Sandridge S, Turk DC, Folmer RL, Frederick EJ, House JW, Jacobson GP, Kinney SE, Martin WH, Nagler SM, Reich GE, Searchfield G, Sweetow R, Vernon JA. The tinnitus functional index: development of a new clinical measure for chronic, intrusive tinnitus. Ear Hear. 2012 Mar-Apr;33(2):153-76. doi: 10.1097/AUD.0b013e31822f67c0. PMID 22156949
- [Background] Li Y, Yang J, Liu J, Wu H. Restudy of malformations of the internal auditory meatus, cochlear nerve canal and cochlear nerve. Eur Arch Otorhinolaryngol. 2015 Jul;272(7):1587-96. doi: 10.1007/s00405-014-2951-4. Epub 2014 Mar 6. PMID 24599597
- [Background] Yan F, Li J, Xian J, Wang Z, Mo L. The cochlear nerve canal and internal auditory canal in children with normal cochlea but cochlear nerve deficiency. Acta Radiol. 2013 Apr 1;54(3):292-8. doi: 10.1258/ar.2012.110596. Epub 2013 Jan 14. PMID 23319716
- [Background] Tahir E, Bajin MD, Atay G, Mocan BO, Sennaroglu L. Bony cochlear nerve canal and internal auditory canal measures predict cochlear nerve status. J Laryngol Otol. 2017 Aug;131(8):676-683. doi: 10.1017/S0022215117001141. Epub 2017 Jun 1. PMID 28566097
- [Background] van der Jagt MA, Brink WM, Versluis MJ, Steens SC, Briaire JJ, Webb AG, Frijns JH, Verbist BM. Visualization of human inner ear anatomy with high-resolution MR imaging at 7T: initial clinical assessment. AJNR Am J Neuroradiol. 2015 Feb;36(2):378-83. doi: 10.3174/ajnr.A4084. Epub 2014 Aug 21. PMID 25147195
- [Background] Peng L, Xiao Y, Liu L, Mao Z, Chen Q, Zhou L, Liao B, Liu A, Wang X. Evaluation of cochlear nerve diameter and cross-sectional area in ANSD patients by 3.0-Tesla MRI. Acta Otolaryngol. 2016 Aug;136(8):792-9. doi: 10.3109/00016489.2016.1159329. Epub 2016 Mar 22. PMID 27003148
- [Background] Kasper JM, Wadhwa V, Scott KM, Rozen S, Xi Y, Chhabra A. SHINKEI--a novel 3D isotropic MR neurography technique: technical advantages over 3DIRTSE-based imaging. Eur Radiol. 2015 Jun;25(6):1672-7. doi: 10.1007/s00330-014-3552-8. Epub 2015 Feb 1. PMID 25638217
- [Background] Zhang H, Schneider T, Wheeler-Kingshott CA, Alexander DC. NODDI: practical in vivo neurite orientation dispersion and density imaging of the human brain. Neuroimage. 2012 Jul 16;61(4):1000-16. doi: 10.1016/j.neuroimage.2012.03.072. Epub 2012 Mar 30. PMID 22484410